CLINICAL TRIAL: NCT01749293
Title: Partially HLA Mismatched (Haploidentical) Allogeneic Bone Marrow Transplantation for Patients With Hematologic Malignancies
Brief Title: Partially HLA Mismatched (Haploidentical) Allogeneic Bone Marrow Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The protocol design is being reconfigured in order to open a new study.
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Pritesh Patel, MD, Faculty, Asst. Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0170
Record Dates: First submitted 2012-11-20; First posted 2012-12-13 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — fludarabine; fludarabine phosphate; Busulfan; Whole-Body Irradiation; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Haploidentical Transplant (Experimental): All subjects will be dosed with pre-transplant Fludarabine (180mg/m2)and Busulfan total AUC 2400 μmol*min/L or 6.4mg/kg. Subjects will then undergo total body irradiation 2Gy. Subjects will undergo haploidentical allogeneic bone marrow transplant, followed by Cyclophosphamide, Tacrolimus and MMF based GVHD prophylaxis.
  Interventions: Procedure: Haploidentical Transplant; Drug: Fludarabine; Drug: Busulfan; Radiation: Total Body Irradiation; Drug: Cyclophosphamide

INTERVENTIONS:
Procedure: Haploidentical Transplant — Subjects will be dosed with pre-transplant Fludarabine (180mg/m2)and Busulfan total AUC 2400 μmol*min/L or 6.4mg/kg. Subjects will then undergo total body irradiation 2Gy. Subjects will undergo haploidentical allogeneic bone marrow transplant, followed by Cyclophosphamide, Tacrolimus and MMF based GVHD prophylaxis.
  Other Names: Mismatched allogeneic bone marrow transplant
Drug: Fludarabine — Subjects in this trial will receive Fludarabine 30 mg/m2 IV QD, adjusted for CrCl from Days -8 through -3.
  Other Names: Fludara
Drug: Busulfan — Subjects in this trial will receive Busulfan total AUC 2400 μmol*min/L or 6.4mg/kg in 4 doses with seizure prophylaxis from Days -6 through -3.
  Other Names: Busulfex; Myleran
Radiation: Total Body Irradiation — Subjects in this trial will receive total body irradiation (2Gy fractionated) from Day -2 or -1.
Drug: Cyclophosphamide — Subjects in this trial will receive Cyclophosphamide 50 mg/kg IV QD on Days 3 and 4 post-transplant.
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune; cytophosphane

SUMMARY:
Allogeneic stem cell transplantation is a potentially curative treatment for patients with many hematologic malignancies (e.g. leukemia, lymphoma, and myeloma with high risk of relapse). This process requires a suitable donor. The best case scenario involves an Human Leukocyte Antigen (HLA) matched sibling donor. However, this type of donor is not always available. Donor registries can provide another source for matched unrelated donors, but this may take valuable time delaying treatment for the transplant recipient. Donor availability remains a significant barrier to the use of allogeneic (from a donor) stem cell transplant. This issue disproportionately affects patients of minority backgrounds. Novel strategies to improve outcomes using alternative donors are desperately needed.

Haploidentical transplants are an alternative which provides a readily available donor in the form of a partially HLA matched family member. This provides for more potential donors and the donors can be selected based on other factors that can play a role in transplant success (e.g. age, gender, KIR alloreactivity). Recent advances in transplant techniques have greatly improved success rates with haploidentical transplants although disease relapse has remained as issue.

This trial aims to provide an alternative transplant option for patients with hematologic malignancies who require bone marrow transplantation but lack an HLA identical donor. The investigational component of this study is the combination of the Fludarabine/ Busulfan/ Total Body Irradiation conditioning regimen and the HLA Haploidentical Transplant with post-transplant Cyclophosphamide.

DETAILED DESCRIPTION:
Allogeneic stem cell transplantation is a potentially curative treatment for patients with hematologic malignancies such as leukemia, lymphoma and myeloma who are at high risk of relapse. As well as the potential to deliver high doses of chemotherapy or radiation this procedure affords the benefit of an immunologic weapon against disease in the form of the graft versus tumor effect.

The major variables affecting the outcome of allogeneic transplant include: patient selection (age and comorbidities); disease status at the time of transplantation (remission vs. active disease); type of donor (HLA matched vs. mismatched or related vs. unrelated); type of conditioning regimen; source of stem cells (bone marrow vs. peripheral blood). Recent advances in the field of stem cell transplant have substantially lowered transplant related morbidity and mortality.

The availability of stem cell transplant as a treatment modality is dependent upon the availability of a suitable donor. Best outcomes are thought to occur in HLA matched sibling donors. The chance of a sibling being HLA matched is approximately 25%. Despite the development of large worldwide donor registries the likelihood of finding an HLA matched unrelated donor is 60-70% at best and drops to 10% in some ethnic minorities. In addition the process of identifying, confirming and harvesting an unrelated donor is cumbersome and time consuming at a time when the patient must proceed immediately to transplant (time from initiation of search to identification of an unrelated donor identification takes a median of 49 days). Therefore the development of alternative sources of hematopoietic stem cells is an area of immense interest to many investigators.

Alternative sources include cord blood and HLA haploidentical donors. Cord blood has been an attractive source permitting immediate availability and possibly a lower rate of graft versus host disease (GVHD). However delay in engraftment, particularly after myeloablative conditioning, remains a significant disadvantage. Haploidentical transplants carry some of the same advantages with virtually all patients having immediate access to a suitable and willing donor in the form of a partially HLA matched family member. Furthermore the number of potential donors allows for donor selection based upon factors such as age, gender, KIR alloreactivity. Finally the donor is readily available for future cellular therapies such as donor lymphocyte infusion.

Early attempts at haploidentical transplantation were hampered by high rates of graft failure and severe graft versus host disease. Recent advances in graft versus host disease prophylaxis with post transplant high dose cyclophosphamide (Cy) have overcome these barriers to a large degree. Published studies have shown that HLA-haploidentical bone marrow transplant (BMT) after non-myeloablative conditioning and using 2 doses of post-transplantation Cy followed by tacrolimus and mycophenolate mofetil (MMF) is a well-tolerated procedure. However, the major cause of treatment failure in this high-risk population was early relapse. As conditioning intensity has been clearly linked to rates of relapse in multiple diseases, it is postulated that utilizing conditioning with higher anti-tumor potential will lead to a lower relapse rate.

Given the advances in GVHD prophylaxis with post-transplantation Cy, reduced intensity conditioning with Fludarabine, Busulfan and total body irradiation combined with high-dose post-transplantation Cy is the platform for this study. The toxicities of this reduced intensity conditioning regimen are not expected to differ substantially from previous data incorporating post-transplantation Cy. However, this regimen may have higher anti-tumor potential resulting in a decreased relapse rate.

ELIGIBILITY:
Inclusion Criteria:

1. First-degree related donor or half-sibling who is at minimum HLA haploidentical
2. Lack of fully matched donor (related or unrelated). Patients with a matched unrelated donor may only be enrolled if they require an urgent transplant. Urgency of transplant will judged by PI and co-investigators.
3. Eligible diagnoses are listed below:

   1. Low-grade non-Hodgkin's lymphoma or plasma cell neoplasm that has progressed during multiagent therapy including follicular lymphoma, Marginal zone (or MALT) lymphoma, lymphoplasmacytic lymphoma / Waldenstrom's macroglobulinemia, Hairy cell leukemia, Small lymphocytic lymphoma (SLL) or chronic lymphocytic leukemia (CLL), Prolymphocytic leukemia, Multiple myeloma and Plasma cell leukemia
   2. Poor-risk SLL or CLL
   3. Aggressive lymphoma that has failed at least one prior regimen of multiagent chemotherapy, and patient is either ineligible for autologous BMT or autologous BMT is not recommended including Hodgkin lymphoma, high grade Follicular lymphoma, Mantle cell lymphoma, Diffuse large B-cell lymphoma, Burkitt's lymphoma/leukemia, Anaplastic large cell lymphoma, Plasmablastic lymphoma, Peripheral T-cell lymphoma
   4. Relapsed or refractory acute leukemias.
   5. Poor-risk acute leukemia in first remission:

   i. Acute myeloid leukemia (AML) with at least one of the following:
   * AML arising from myelodysplastic syndrome (MDS) or a myeloproliferative disorder
   * Presence of FLT3 internal tandem duplications
   * Poor-risk cytogenetics

   ii. Acute lymphoblastic leukemia and/or lymphoma (ALL) with at least one of the following:
   * Poor risk cytogenetics
   * Primary refractory disease

   iii. Biphenotypic leukemia

   f. MDS with at least one of the following poor-risk features: i. Poor-risk cytogenetics ii. Int-2 or high IPSS score iii. Treatment-related MDS iv. MDS diagnosed before age 21 years v. Progression on or lack of response to standard hypomethylator therapy vi. Life-threatening cytopenias

   g. Imatinib-refractory chronic myelogenous leukemia (CML) in accelerated or chronic phase

   h. Philadelphia chromosome negative myeloproliferative neoplasm

   i. Chronic myelomonocytic leukemia

5. Adequate end-organ function as measured by:

1. Left ventricular ejection fraction ≥ 35%
2. Bilirubin ≤ 3.0 mg/dL and ALT and AST < 5 x ULN
3. FEV1 and FVC > 40% of predicted

   6. Karnofsky score > 60

   7. Lack of recipient anti-donor HLA antibody

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-08-30 (Actual); Primary Completion 2014-05-15 (Actual); Study Completion 2014-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pritesh Patel, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Cancer Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Haploidentical Transplant
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Haploidentical Transplant: All subjects will be dosed with pre-transplant Fludarabine (180mg/m2)and Busulfan total AUC 2400 μmol*min/L or 6.4mg/kg. Subjects will then undergo total body irradiation 2Gy. Subjects will undergo haploidentical allogeneic bone marrow transplant, followed by Cyclophosphamide, Tacrolimus and MMF based GVHD prophylaxis.
  Fludarabine: Subjects in this trial will receive Fludarabine 30 mg/m2 IV QD, adjusted for CrCl from Days -8 through -3.
  Busulfan: Subjects in this trial will receive Busulfan total AUC 2400 μmol*min/L or 6.4mg/kg in 4 doses with seizure prophylaxis from Days -6 through -3.
  Total Body Irradiation: Subjects in this trial
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.8 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Engrafted and the Number of Participants That Had Full Donor Chimerism at Day 60
Description: To estimate the number of participants that had engraftment rates and the number of participants that had full donor chimerism at Day 60 in patients undergoing an HLA haploidentical stem cell transplant with post transplant high dose cyclophosphamide.
Time Frame: Up to Day 60 post-transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Number of Participants That Had an Overall Survival Rate
Description: To estimate the number of participants that had an overall survival (OS) rate
Time Frame: Up to one year post-transplant.
Measure: Count of Participants; unit: Participants
Groups:
- Haploidentical Transplant: All subjects will be dosed with pre-transplant Fludarabine (180mg/m2)and Busulfan total AUC 2400 μmol*min/L or 6.4mg/kg. Subjects will then undergo total body irradiation 2Gy. Subjects will undergo haploidentical allogeneic bone marrow transplant, followed by Cyclophosphamide, Tacrolimus and MMF based GVHD prophylaxis.
  Haploidentical Transplant: Subjects will be dosed with pre-transplant Fludarabine (180mg/m2)and Busulfan total AUC 2400 μmol*min/L or 6.4mg/kg. Subjects will then undergo total body irradiation 2Gy. Subjects will undergo haploidentical allogeneic bone marrow transplant, followed by Cyclophosphamide, Tacrolimus and MMF based GVHD prophylaxis.
  Fludarabine: Subjects in this trial will receive Fludarabine 30 mg/m2 IV QD, adjusted for CrCl from Days -8 through -3.
  Busulfan: Subjects in this trial will receive Busulfan total AUC 2400 μmol*min/L or 6.4mg/kg in 4 doses with seizure prophylaxis from Days -6 through -3.
  Total Body Irradiation: Subjects in this trial
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 3
Participants | 1

3. Secondary Outcome: Number of Participants That Had an Event Free Survival Rate
Description: To estimate the number of participants who had an event free survival rate
Time Frame: Up to 1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Haploidentical Transplant
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haploidentical Transplant (N=3)
Serious (Cardiac disorders) | 1 (1) — Subject became short of breath and tachycardic to 180 per ECG, B/P60/40 and O2 saturation 74%. Subject administered adenosine IV and his heart rate and shortness of breath improved

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No